

## **Informed Consent Form**

## NCT05683158

| Research Project Title: | Compensatory Kinematic Movements in Various Directions After Stroke |
|---|---|
| IRB Approval Number: | UNISTIRB-22-43-A |

Do you consent to the secondary use of your research data (samples) or specimens for purp oses other than those stated in this informed consent form?

| Without additional consent, the data (samples) will be used in a state that includes personally identifiable information |
|---|
| Without additional consent, the personally identifiable information in the data (samples) will be encoded, allowing for the possibility of tracing and identifying the research participants |
| Without additional consent, the personally identifiable information in the data (samples) will be completely removed and utilized in a state where individual identification is not possible |
| If the data (samples) are to be used for a different type of research, please proceed with obtaining my additional informed consent before proceeding |
| I agree. I confirm that you do not consent to the use of the data (samples) for purposes other than those stated in the informed consent |

I hereby confirm that I have no relationships that could influence my decision to participate in the research, between myself, the researchers, and UNIST

I affirm that I have received an explanation of this consent form from the research personnel, have personally read and understood it, and have received satisfactory answers to all my questions. I voluntarily and without any coercion sign this consent form to confirm my participation in this research

## (The date and signature must be handwritten)

| Participant | (Name) | (Signature) | (The date) |
|---|---|---|---|
| Legal Guardian (If necessary) | (Name) | (Signature) | (The date) |
| | (Relationship with legal guardian) | | |



## 심의서식6 (version 4.0, 2022.07)

| Applicant (If necessary) | (Name) | (Signature) | (The date) |
|--------------------------|--------|-------------|------------|
| Principal Investigator | (Name) | (Signature) | (The date) |
| Co-Investigator | (Name) | (Signature) | (The date) |

This research will only utilize consent forms that have been reviewed and approved by the UNIST IRB(Institutional Review Board)